CLINICAL TRIAL: NCT02335060
Title: Effect of N-acetylcysteine on the Acute Cognitive Effects of Delta-9-Tetrahydrocannabinol
Brief Title: N-acetylcysteine Effects on Tetrahydrocannabinol
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Feasibility pilot was completed
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Mohini Ranganathan, Principal Investigator, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1402013406
Record Dates: First submitted 2015-01-05; First posted 2015-01-09 (Estimated); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Healthy
Keywords: cannabis; Marijuana; THC; N-acetylcysteine; Psychotic Disorders
MeSH Terms: conditions — Marijuana Abuse; Psychotic Disorders | interventions — Dronabinol; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Active N-acetylcysteine and Active Delta-9-THC (Experimental)
  Interventions: Drug: Delta-9-THC; Drug: N-acetylcysteine
- Placebo and Active Delta-9-THC (Placebo Comparator)
  Interventions: Drug: Delta-9-THC; Drug: Placebo
- Active N-acetylcysteine and Placebo (Experimental)
  Interventions: Drug: N-acetylcysteine; Drug: Placebo
- Placebo and Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Delta-9-THC — Active Delta-9-THC (0.036mg/Kg) given intravenously.
  Arms: Active N-acetylcysteine and Active Delta-9-THC; Placebo and Active Delta-9-THC
Drug: N-acetylcysteine — A pill given orally.
  Arms: Active N-acetylcysteine and Active Delta-9-THC; Active N-acetylcysteine and Placebo
Drug: Placebo — Placebo (about a quarter spoon of alcohol with no THC) given intravenously.
  Arms: Active N-acetylcysteine and Placebo; Placebo and Placebo
Drug: Placebo — Placebo "sugar" pill given orally with no N-acetylcysteine.
  Arms: Placebo and Active Delta-9-THC; Placebo and Placebo

SUMMARY:
The overall purpose of this study is to examine the effect of N-acetylcysteine (NAC) on the acute effects of Delta-9-tetrahydrocannabinol (THC). This will be tested by pretreating healthy individuals with NAC and then assessing their responses to THC.

ELIGIBILITY:
Inclusion Criteria:

* Exposed to Cannabis at least once in lifetime

Exclusion Criteria:

* Cannabis Naive
* Individuals with a documented allergy to N-acetylcysteine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2014-05-02 (Actual); Primary Completion 2014-09-16 (Actual); Study Completion 2014-09-16 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Symptom Scale for Schizophrenia (PANSS) | -30 minutes from administration of THC
  Positive, negative, and general symptoms will be assessed using the positive, negative, and general symptom subscales of the PANSS
Positive and Negative Symptom Scale for Schizophrenia (PANSS) | +15 minutes from administration of THC
  Positive, negative, and general symptoms will be assessed using the positive, negative, and general symptom subscales of the PANSS
Positive and Negative Symptom Scale for Schizophrenia (PANSS) | +90 minutes from administration of THC
  Positive, negative, and general symptoms will be assessed using the positive, negative, and general symptom subscales of the PANSS
Positive and Negative Symptom Scale for Schizophrenia (PANSS) | +240 minutes from administration of THC
  Positive, negative, and general symptoms will be assessed using the positive, negative, and general symptom subscales of the PANSS
Positive and Negative Symptom Scale for Schizophrenia (PANSS) | -60 minutes from administration of THC
  Positive, negative, and general symptoms will be assessed using the positive, negative, and general symptom subscales of the PANSS

SECONDARY OUTCOMES:
Clinician Administered Dissociative Symptoms Scale (CADSS) | -60min, -30min, +15min, +90min, +240min from administration of THC
  Perceptual alterations will be measured using the CADSS. This is a scale consisting of 19 self-reported items and 8 clinician-rated items. The scale captures alterations in environmental/time/body perception, feelings of unreality, and memory impairment.
Visual Analog Scale (VAS) | -60min, -30min, +15min, +90min, +240min from administration of THC
  Feeling states associated with cannabis intoxication will be measured using a self-reported visual analog scale of feeling states associated with cannabis effects (ex: "high," "calm," "anxious"). Subjects will be asked to score the perceived intensity of these feeling states at that moment on a 11mm line. These data will be captured to validate that the experiment is relevant to cannabis effects.
Cognitive Test Battery | +20min from administration of THC
  Several computer tasks will be administered in order to evaluate the effects of cannabis on recognition memory, working memory, and attention. The battery consists of four computer tasks that lasts no longer than 20 minutes in total.
Hopkins Verbal Learning Test (HVLT) | +20min from administration of THC
  The HVLT is a 12 word list that is semantically organized. The task consists of 5 trials and a different version of the HVLT will be administered on each test day.
Psychotomimetic States Inventory (PSI) | -60min, -30min, +240min from administration of THC
  The PSI is a measure of drug induced psychotomimetic states. This self-reported scale consists of 28 items rated 0 (not at all) to 3 (extremely) and will facilitate the characterization of a wide range of dissociative/hallucinatory phenomena as well as cognitive disorganization associated with the administration of THC.

CONTACTS AND LOCATIONS:
Overall Officials: Mohini Ranganathan, MD, Principal Investigator — Yale University Medical School
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States